CLINICAL TRIAL: NCT01839513
Title: Prediction of Hemodynamic Reactivity During Desflurane/Remifentanil General Anesthesia Using Analgesia/Nociception Index (ANI)
Brief Title: Prediction of Hemodynamic Reactivity During General Anesthesia Using Analgesia/Nociception Index (ANI)
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Emmanuel Boselli, MD, PhD, Hôpital Edouard Herriot
Other Study IDs: CPP 2013-021B
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Anesthesia
Keywords: Analgesia/nociception index; Desflurane; Remifentanil; Orthopedic surgery; Ear-nose-throat surgery; Hemodynamic reactivity
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to evaluate the performance of Analgesia/Nociception Index for the prediction of hemodynamic reactivity in adult patients undergoing ear-nose-throat or lower limb orthopedic surgery on desflurane/remifentanil general anesthesia.

DETAILED DESCRIPTION:
Measurement of analgesia/nociception index at different time points during procedure and assessment of analgesia/nociception index to predict hemodynamic reactivity by building receiver observer's characteristic curve.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Ear-nose-throat or lower limb surgery
* General anesthesia using desflurane and remifentanil

Exclusion Criteria:

* Age <18 yrs or >75 yrs
* Arrythmia
* Preoperative use of B-blockers
* Administration of anticholinergic drugs or neuromuscular blockade reversal in the 20 previous minutes
* Psychiatric diseases
* Autonomic nervous system disorders (epilepsy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients underoing ear-nose-throat or orthopedic lower limb surgery performed on desflurane/remifentanil general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in heart rate and/or systolic blood pressure by more than 20% within 5 minutes | Before induction of anesthesia, 1 min after incision, at steady-state anesthesia during procedure (an expected average of 30 min) and at arousal from general anesthesia in the end of procedure (an expected average of 60 min)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Boselli, MD, PhD, Study Director — Hôpital Edourd Herriot; Bernard Allaouchiche, MD, PhD, Study Chair — Hôpital Edouard Herriot
Locations (1):
- Hôpital Édouard Herriot, HCL, Lyon, Rhône, France

REFERENCES:
- [Background] Boselli E, Daniela-Ionescu M, Begou G, Bouvet L, Dabouz R, Magnin C, Allaouchiche B. Prospective observational study of the non-invasive assessment of immediate postoperative pain using the analgesia/nociception index (ANI). Br J Anaesth. 2013 Sep;111(3):453-9. doi: 10.1093/bja/aet110. Epub 2013 Apr 16. PMID 23592690